CLINICAL TRIAL: NCT01107392
Title: Safety and Efficacy of Botulinum Toxin Type A to Treat Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-100
Record Dates: First submitted 2010-04-16; First posted 2010-04-21 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin Type A (Experimental): botulinum toxin Type A total dose of 200U equally divided and administered to each lateral prostatic lobe.
  Interventions: Drug: botulinum toxin Type A
- Placebo (Normal saline) (Placebo Comparator): Placebo (Normal saline) equally divided and administered to each lateral prostatic lobe.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: botulinum toxin Type A — botulinum toxin Type A total dose of 200U equally divided and administered to each lateral prostatic lobe.
  Other Names: BOTOX®; onabotulinumtoxinA
  Arms: botulinum toxin Type A
Drug: Normal saline — Placebo (Normal saline) equally divided and administered to each lateral prostatic lobe.
  Arms: Placebo (Normal saline)

SUMMARY:
This study will evaluate the safety and efficacy of intraprostatic administration of botulinum toxin Type A (BOTOX®) compared with placebo to treat urinary tract symptoms due to benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical enlargement of the prostate gland
* Body weight ≥ 50 kg or 110 lbs

Exclusion Criteria:

* History of chronic prostatitis
* History of two or more urinary tract infections in the past year or one in the last 6 months
* History of bladder stones
* History of previous prostate surgery
* History of bladder cancer or prostate cancer
* Any previous or current usage of botulinum toxin therapy of any serotype for any urological condition
* Botulinum toxin therapy of any serotype for any non-urological condition or usage (e.g., cosmetic) during the previous 12 weeks prior to study entry

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2012-03-16 (Actual); Study Completion 2012-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (8):
- Newport Beach, California, United States
- Surrey, British Columbia, Canada
- Prague, Czechia
- Paris, France
- Munich, Germany
- Manila, Philippines
- Poznan, Poland
- Seoul, South Korea

REFERENCES:
- [Background] McVary KT, Roehrborn CG, Chartier-Kastler E, Efros M, Bugarin D, Chen R, Patel A, Haag-Molkenteller C. A multicenter, randomized, double-blind, placebo controlled study of onabotulinumtoxinA 200 U to treat lower urinary tract symptoms in men with benign prostatic hyperplasia. J Urol. 2014 Jul;192(1):150-6. doi: 10.1016/j.juro.2014.02.004. Epub 2014 Feb 7. PMID 24508634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Started | 158 | 157
Completed | 153 | 154
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Personal Reasons | 2 | 3
Not completed — Administrative decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 Years | 89 (8.19) | 79 (8.12) | 168
  > 65 Years | 69 | 78 | 147
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 158 | 157 | 315

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total International Prostate Symptom Score (IPSS) at Week 12
Description: IPSS is a disease-specific outcome measure based on the American Urological Association Symptom Index. The questionnaire consisted of seven items. The patient evaluated their urinary symptoms (incomplete emptying, frequency, hesitancy, urgency, weak stream, straining, and nocturia) during the previous 4 weeks. The total symptom score ranged from 0 (no symptoms) to 35 (most severe symptoms). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Modified Intent-to-treat population included all randomized and treated participants with at least one post-baseline IPSS measurement.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 156 | 157
Score on a scale
  Baseline | 21.8 (4.90) | 21.5 (4.56)
  Change from Baseline at Week 12 | -6.3 (6.61) | -5.6 (5.86)

2. Secondary Outcome: Change From Baseline in the Total International Prostate Symptom Score (IPSS)
Description: as for outcome 1
Time Frame: Baseline, Week 6, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 156 | 157
Score on a scale
  Baseline | 21.8 (4.90) | 21.5 (4.56)
  Change from Baseline at Week 6 (n=156,156) | -5.4 (5.84) | -5.3 (5.27)
  Change from Baseline at Week 24 (n=152,154) | -6.3 (6.43) | -6.0 (5.79)

3. Secondary Outcome: Change From Baseline in Peak Urine Flow Rate
Description: Urinary flow was determined by uroflowmetry measured in milliliters/second (mL/sec). An increase from Baseline indicated improvement.
Time Frame: Baseline, Weeks 6, 12 and 24
Population: Modified Intent-to-treat population included all randomized and treated participants with at least one post-baseline IPSS measurement with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 154 | 156
mL/sec
  Baseline | 8.0 (2.52) | 8.0 (2.86)
  Change from Baseline at Week 6 (n=138,136) | 2.5 (4.97) | 1.2 (3.40)
  Change from Baseline at Week 12 (n=143,147) | 2.5 (5.24) | 1.7 (4.38)
  Change from Baseline at Week 24 (n=140,149) | 2.5 (4.97) | 1.9 (4.32)

4. Secondary Outcome: Duration of Effect
Description: Duration of effect was calculated from the time of the first follow-up visit with a ≥ 4-point reduction from Baseline in IPSS to the next visit when the IPSS change from Baseline was < 4-points.
Time Frame: 24 Weeks
Population: Modified Intent-to-treat population included all randomized and treated patients with at least one post-baseline IPSS measurement. Only patients with at least a 4-point reduction from Baseline in total IPSS were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 123 | 120
Weeks | 20.9 [18.6 to 20.9] | 20.6 [20.1 to NA] — Not estimable.

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 5/158 | 8/157
Other Adverse Events (participants affected / at risk) | 42/158 | 44/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=158) | Placebo (Normal Saline) (N=157)
Retinal detachment (Eye disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=158) | Placebo (Normal Saline) (N=157)
Prostatic specific antigen increased (Investigations) | 6 | 10
Haematuria (Renal and urinary disorders) | 23 | 18
Haematospermia (Reproductive system and breast disorders) | 13 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.